CLINICAL TRIAL: NCT01143883
Title: A Randomized Controlled Clinical Trial Evaluating the Efficacy of Silverlon® in Preventing Surgical Site Infection Following Colorectal Surgery
Brief Title: Study Looking at the Effect of Silverlon on Post Operative Wound Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jorge Marcet (Other)
Responsible Party: Sponsor-Investigator, Jorge Marcet, Professor, Department of Surgery, University of South Florida
Organization: University of South Florida (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Silverlon 108010
Record Dates: First submitted 2010-03-24; First posted 2010-06-14 (Estimated); Results first posted 2013-06-13 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Infections; Surgery
Keywords: All patients undergoing a colorectal resection; surgical site infections
MeSH Terms: conditions — Infections; Surgical Wound Infection | interventions — silverlon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Silverlon Dressing (Experimental): The Silverlon(Cura Surgical, Geneva, IL) dressing is applied to the surgical wound postoperatively. This dressing is coated with silver nylon.
  Interventions: Other: Silverlon
- Standard of Care Dressing (Active Comparator): The standard plain gauze is used to dress the wound postoperatively
  Interventions: Other: Standard of Care Dressing

INTERVENTIONS:
Other: Silverlon — Silverlon dressings are gauze impregnated with silver ions
  Arms: Silverlon Dressing
Other: Standard of Care Dressing — Standard dry gauze dressing
  Arms: Standard of Care Dressing

SUMMARY:
This clinical study is a prospective, randomized, controlled trial of patients undergoing elective colorectal surgical procedures that receive an abdominal skin incision of at least 6 cm. Treatment with Silverlon® will be compared to standard postoperative dressings of 4x4 Gauze and paper tape. Patients will be randomized with a 1:1 treatment allocation ratio to receive either 1) Silverlon® or 2) standard postsurgical dressing. Neither the Investigators nor the participants will be blinded to the treatment modality after randomization.

Silver has long been known to have antimicrobial properties. It interacts with structural proteins and DNA, inhibiting bacterial replication and causing fatal structural changes within the cell wall. It has broad antimicrobial activities and unlike antibiotics, it is rarely associated with microbial resistance. Silverlon® is a silver-nylon dressing specifically designed for surgical wounds to prevent the development of surgical site infections. It is an easy to use product with no known microbial resistance or adverse effects. The efficacy of Silverlon® in preventing surgical site infections has been shown in several retrospective studies but as of yet has not been tested in a prospective fashion. The objective of this study is to perform a prospective, randomized, clinical trial directly comparing the incidence of surgical site infections in patients treated with Silverlon® to standard postoperative dressing following elective colorectal surgery

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing elective colorectal surgery by a trained colorectal surgeon with an abdominal skin incision of at least 3 cm
2. Patients that are willing and able to comply with the requirements of the protocol including follow-up requirements
3. Patients willing and able to sign a study specific informed consent

Exclusion Criteria:

1. Patients that fail to meet the skin incision size criteria
2. Patients with a known allergy to silver
3. Patients less than 18 years of age
4. Any contraindication to undergoing a surgical procedure under general anesthesia
5. Patients with preoperative evidence of a current abdominal wall infection/surgical site infection from a previous laparotomy/laparoscopy
6. Patients that have received antibiotic therapy within the week prior to surgery
7. Patients with preoperative evaluation suggestive of an intra-abdominal process that would preclude full closure of the skin
8. Patients with a previously placed anterior abdominal wall mesh that is not planned to be completely removed during the planned procedure
9. Women who are pregnant or breast feeding or are considering becoming pregnant during the follow-up period
10. Mental incompetence as determined by the Investigator which would affect participation in the study
11. Concurrently participating in any other investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tampa General Hospital and University of South Florida Medical Clinics, Tampa, Florida, United States

REFERENCES:
- [Derived] Krieger BR, Davis DM, Sanchez JE, Mateka JJ, Nfonsam VN, Frattini JC, Marcet JE. The use of silver nylon in preventing surgical site infections following colon and rectal surgery. Dis Colon Rectum. 2011 Aug;54(8):1014-9. doi: 10.1097/DCR.0b013e31821c495d. PMID 21730792

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All 110 patients were consented for this study during their pre-operative visit.
Period: Overall Study
Arm/Group | Silverlon Dressing | Standard of Care Dressing
Started | 55 | 55
Completed | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Silverlon Dressing; Standard of Care Dressing: 55
- Total: Total of all reporting groups
Arm/Group | Silverlon Dressing | Standard of Care Dressing | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 3 | 3
  Between 18 and 65 years | 45 | 4 | 49
  >=65 years | 10 | 48 | 58
Age Continuous [Mean (Standard Deviation); unit: years] | 62 (15.6) | 58 (11.1) | 60 (13.7)
Gender [Number; unit: participants]
  Female | 27 | 28 | 55
  Male | 28 | 26 | 54
Region of Enrollment [Number; unit: participants]
  United States | 55 | 55 | 110

OUTCOME MEASURES:

1. Primary Outcome: Surgical Site Infection
Description: We will monitor the incision from the day of surgery to post operative day 30 to determine if the incision needs antibiotics.
Time Frame: Day of surgery up to 30 days post operatively
Population: The number of participants analyzed was based on the number who received treatment according to their randomized group and were treated according to study protocol
Measure: Number; unit: percentage of participants with SSI
Arm/Group | Silverlon Dressing | Standard of Care Dressing
Number analyzed (Participants) | 55 | 54
percentage of participants with SSI | 13 | 33

ADVERSE EVENTS:
Arm/Group | Silverlon Dressing | Standard of Care Dressing
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 1/55 | 0/55
OTHER ADVERSE EVENTS (reported when occurring in more than 1.82% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Silverlon Dressing (N=55) | Standard of Care Dressing (N=55)
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 — Rash resolved after dressing removed

LIMITATIONS AND CAVEATS:
Members of the surgical team were not blinded to the treatment group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No